CLINICAL TRIAL: NCT02194608
Title: A Randomized Clinical Trial on Home Telemonitoring for the Management of Metabolic and Cardiovascular Risk in Individuals With Type 2 Diabetes
Brief Title: Telemonitoring System Study in Participants With Type 2 Diabetes Mellitus (MK-0000-347)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0000-347; LCE#40378 (Other: Merck)
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedicine system (Experimental): Participants will self-test blood glucose level, weight, and blood pressure and results will be uploaded and transmitted directly via a hometelehealth system to a central location (HUB). Blood draws will be administered at baseline and follow-up visits.
  Interventions: Device: Home telehealth system
- Usual care (No Intervention): Participants will self-record their blood glucose levels, blood pressure and weight in a diary. Blood draws will be administered at baseline and follow-up visits.

INTERVENTIONS:
Device: Home telehealth system — Participants will receive a weighing machine, glucometer, and a sphygmomanometer connected through a Bluetooth system from their home to the Telehealth center via a HUB.
  Arms: Telemedicine system

SUMMARY:
The primary goal is to evaluate whether a home telehealth system that enables the participant to monitor their body weight, blood glucose values and blood pressure values, associated with remote educational support and feedback to the general practitioner, can improve metabolic control and overall cardiovascular risk in individuals with type 2 diabetes mellitus (T2DM), as compared to usual practice.

ELIGIBILITY:
Inclusion Criteria:

* has type 2 diabetes
* treated with oral agents in monotherapy or combined therapy ± basal insulin
* previously educated to self-monitoring blood glucose (SMBG) use

Exclusion Criteria:

* has type 2 diabetes non-pharmacologically treated
* has type 2 diabetes treated with multiple daily injections of insulin
* is unable to use the telemedicine system
* pregnancy
* has major cardiovascular, cerebrovascular, or peripheral vascular event in the last 6 months
* has any disease or condition, including alcohol or drugs abuse, that may interfere with study completion

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in blood glucose level | Baseline and 12 months
Change from baseline in blood pressure | Baseline and 12 months
Change from baseline in body mass index | Baseline and 12 months

SECONDARY OUTCOMES:
Percentage of participants who achieved hemoglobin A1c (HbA1c) <7.0% | Up to 12 months
Percentage of participants who achieved blood pressure <130/80 mmHg | Up to 12 months
Percentage of participants who achieved low-density lipoprotein (LDL) cholesterol <100 mg/dL | Up to 12 months
Percentage of participants requiring therapy modifications | Up to 12 months
Change from baseline in total cholesterol | Baseline, 6 months, and 12 months
Change from baseline in high-density lipoprotein (HDL) cholesterol | Baseline, 6 months, and 12 months
Change from baseline in LDL cholesterol | Baseline, 6 months, and 12 months
Change from baseline in triglycerides | Baseline, 6 months, and 12 months
Change from baseline in cardiovascular risk score | Baseline, 6 months, and 12 months
Number of emergency room visits and hospital admissions | Up to 12 months
Number of office visits and home visits | Up to 12 months
Change from baseline in the number and doses of drugs for treatment of diabetes | Baseline and 12 months
Change from baseline in the number and doses of drugs for treatment of hypertension | Baseline and 12 months
Change from baseline in the number and doses of drugs for treatment of dyslipidemia | Baseline and 12 months
Participant overall satisfaction level | Up to 12 months
Participant compliance with protocol-provided devices | Up to 12 months
Number of participants who experienced hypoglycemia | Up to 12 months
Number of hypoglycemic episodes | Up to 12 months
Number of participants who experienced severe/symptomatic hypoglycemia | Up to 12 months
Number of severe/symptomatic hypoglycemic episodes | Up to 12 months

REFERENCES:
- [Derived] Nicolucci A, Cercone S, Chiriatti A, Muscas F, Gensini G. A Randomized Trial on Home Telemonitoring for the Management of Metabolic and Cardiovascular Risk in Patients with Type 2 Diabetes. Diabetes Technol Ther. 2015 Aug;17(8):563-70. doi: 10.1089/dia.2014.0355. Epub 2015 Jul 8. PMID 26154338